CLINICAL TRIAL: NCT07317882
Title: Effectiveness of a Telematic Educational Intervention in Improving Self-care Levels in Patients With Heart Failure
Brief Title: Telematic Educational Intervention in Patients With Heart Failure.
Acronym: TEACH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Jose Santi Cano (Other)
Responsible Party: Sponsor-Investigator, Maria Jose Santi Cano, Doctor of Medicine, University of Cadiz
Organization: University of Cadiz (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI-25-07-2024
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Heart Failure Patients
Keywords: Heart failure; digital health; self care
MeSH Terms: conditions — Heart Failure | interventions — Digital Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital health (Experimental)
  Interventions: Behavioral: Digital health
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Digital health — Education through mHealth
  Arms: Digital health

SUMMARY:
Background: Heart Failure (HF) is one of the most prevalent pathologies in Western countries, representing a significant percentage of their healthcare expenditure. Much of the success of specialised programmes for the control and treatment of this pathology is achieved within Heart Failure Units. These programmes are based on enhancing patients' capacity to perform effective self-care. Self-care in heart failure involves several aspects: maintaining healthy lifestyle habits, monitoring signs and symptoms of decompensation, controlling blood pressure, heart rate, and body weight, and the ability to manage potential decompensations either autonomously or by seeking available healthcare services.

Heart failure units carry out structured therapeutic education for these patients through individualized, face-to-face educational interventions upon admission to the unit, placing special emphasis on training patients and their caregivers in effective self-care. However, studies show that the level of self-care among HF patients remains low. Furthermore, the new healthcare reality following the pandemic situation necessitates the search for strategies that facilitate better time management while improving the self-care capacity of HF patients. Within this clinical context, it is necessary to seek alternatives that allow for the provision of adequate quality of care while overcoming the obstacles imposed by the current situation.

Objective: The objective of the study is to evaluate the effectiveness of a telematics-based educational intervention, in addition to the standard standardised educational intervention, in self-care in patients in the Heart Failure Unit six months after admission.

Methodology: A randomised clinical trial design with parallel groups (intervention and control) will be applied. The study sample, consisting of 50 patients in each group, will be recruited from patients treated in the Heart Failure Unit of the University Hospital. All patients and their caregivers (if applicable) in both groups will receive the same individualised educational intervention. The patients assigned to the intervention group will also receive a telematics-based educational intervention through video call through the WhatsApp messaging application three months after the initial face-to-face intervention.

The study variables will include sociodemographic and physiological data, adherence to pharmacological treatment, immunisations, dietary assessment, physical exercise assessment, number and management of decompensations, self-care levels and quality of life. After six months in the heart failure unit, all patients in both groups will be reassessed using the same instruments and the statistical differences between the groups will be analysed. The primary outcome variable will be the level of self-care, measured by the European Heart Failure Self-care Behaviour Scale.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age.
* Clinical diagnosis of heart failure class II, III and IV.
* Ejection fraction less than or equal to 35%.
* Those who have a smartphone that allows video calls.

Exclusion Criteria:

* Patients with impaired cognitive ability, meaning they cannot follow basic self-care and education guidelines.
* Patients with acute heart failure that can be resolved by treating the underlying cause.
* Patients with high comorbidity, where non-cardiac conditions pose a greater risk and have a worse prognosis than heart failure itself.
* Patients enrolled in any other clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-03-07 (Estimated); Study Completion 2026-06-07 (Estimated)

PRIMARY OUTCOMES:
European Heart Failure Self-Care Behaviour Scale | From enrollment to the end of intervention at 6 months
  It consists of a 12-item self-administered questionnaire that addresses different aspects of patient self-care. It is scored using a Likert scale from 1 (strongly agree/always) to 5 (strongly disagree/never). This allows for the classification of the overall self-care level within the following ranges: low (44-60), medium (28-43), and high (12-27).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Jerez, Cadiz, Cádiz, Spain

IPD SHARING:
Plan to Share IPD: Yes